CLINICAL TRIAL: NCT07118345
Title: Early Prophylactic Decompressive Hemicraniectomy Following Endovascular Therapy in Large Hemispheric Infarct Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IAT-EPIC
Record Dates: First submitted 2025-06-29; First posted 2025-08-12 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-08

CONDITIONS: Stroke, Ischemic; Cerebral Edema
Keywords: Acute Ischemic Stroke; Endovascular Thrombectomy; Cerebral Edema; Hemicraniectomy
MeSH Terms: conditions — Ischemic Stroke; Brain Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Early prophylactic decompressive hemicraniectomy
  Interventions: Procedure: Early prophylactic decompressive hemicraniectomy
- Control group (No Intervention): Standard medical treatment (with or without rescue decompressive craniectomy if needed).

INTERVENTIONS:
Procedure: Early prophylactic decompressive hemicraniectomy — Early prophylactic decompressive hemicraniectomy (decompressive hemicraniectomy is required to initiate within 6 hours after completion of mechanical thrombectomy and within 4 hours after randomization).
  Arms: Experimental group

SUMMARY:
Early Decompressive Hemicraniectomy for High-Risk Large Ischemic Core Stroke Post-EVTAcute Ischemic Stroke (AIS), particularly Anterior Circulation Large Vessel Occlusion (LVO), is a major cause of global disability and death. While endovascular thrombectomy (EVT) is the standard first-line treatment for LVO, outcomes remain poor in patients with large ischemic cores (ASPECTS ≤5). Despite high recanalization rates (>90%), only 14-30% achieve functional independence (mRS 0-2) at 90 days, with 33-50% dead or severely disabled (mRS 5-6). Outcomes worsen dramatically with larger core volumes (e.g., only 4.4% functional independence with cores ≥150mL in SELECT2).A critical complication is Malignant Cerebral Edema (MCE), affecting ~50% of large-core patients post-EVT. MCE triggers a vicious cycle of rising intracranial pressure, reduced perfusion, and brain herniation. It drastically worsens prognosis: functional independence rates plummet (13.3% vs 51.2% without MCE), mortality significantly increases (OR=7.96, p=0.001), and functional outcomes deteriorate (OR=7.83, p=0.008). Strong predictors include low ASPECTS (<7) and large infarct volume.Decompressive Hemicraniectomy (DHC) is a life-saving intervention for MCE. Landmark trials (DESTINY, DECIMAL, HAMLET) and their meta-analysis show DHC within 24 hours in patients aged 18-60 significantly increases 12-month survival (78% vs 29%, ARR 50%) and rates of ambulatory independence (mRS ≤3: 43% vs 21%, ARR 23%). DESTINY II confirmed benefit in patients >60, improving functional outcomes (mRS 0-4: 38% vs 16%). Guidelines endorse DHC for large infarcts with deterioration.However, significant challenges persist:

DHC is Underutilized: Despite evidence, clinical adoption remains low.Rescue DHC Fails to Improve Outcomes in Post-EVT MCE: Studies report poor functional outcomes (only 20% mRS 0-2) and high mortality (48.6%) with standard medical therapy (SMT) plus rescue DHC after MCE develops. Retrospective data confirms worse outcomes in these patients (mRS 0-2: 16.4% vs 50%; mortality: 46.5% vs 20%) compared to those without MCE. Crucially, rescue DHC itself fails to improve prognosis once MCE is established (mRS 5-6: 64% vs 57.7%; mortality: 48% vs 46.2%).High-Risk Identification: Patients defined as high-risk for MCE (ASPECTS 3-5 + NIHSS≥30 or ASPECTS≤2) have significantly worse 90-day outcomes (mRS 0-2: 23.2% vs 44.6%; mortality: 44% vs 22.7%).Timing is Critical: Rescue DHC is often performed too late, after irreversible neurological damage occurs. Early/Prophylactic DHC, performed before significant edema and herniation develop, offers a potential pathophysiological advantage. It may:Improve cerebral perfusion pressure earlier. Reduce mass effect and edema progression. Mitigate secondary injury (e.g., reduce oxygen-free radicals, excitatory amino acids).Potentially break the ischemic-edema-herniation cycle sooner.Rationale for the Study: While DHC is effective for established MCE in non-EVT contexts and rescue DHC post-EVT is ineffective, high-quality evidence for early prophylactic DHC in high-risk large-core patients after successful EVT is lacking. Current guidelines do not address this specific, high-risk population where MCE incidence is ~50% and outcomes are dismal despite recanalization.

Study Aim: This trial will evaluate the efficacy and safety of early prophylactic decompressive hemicraniectomy compared to standard medical treatment (which includes rescue DHC if MCE develops) in AIS-LVO patients at high risk of MCE (defined by ASPECTS and NIHSS criteria) following successful EVT. The goal is to determine if proactive intervention can improve functional outcomes and reduce mortality in this critically ill population where current strategies fail.

ELIGIBILITY:
1. Premorbid mRS ≤1;
2. Time from symptom onset to puncture ≤24 hours; including wake-up stroke and unwitnessed stroke. The time at which symptoms began was defined as the "Last Known Well" (LKW).

3.18 to 75 years of age; 4.Internal carotid artery (ICA) or middle cerebral artery (MCA)-M1 occlusion confirmed by computed tomographic angiography (CTA)/ magnetic resonance angiography (MRA)/ digital subtraction angiography (DSA). Patients with involvement of ipsilateral anterior cerebral artery (ACA), MCA or embryonal posterior cerebral artery (PCA) are eligible for inclusion.

5.NIHSS1a ≥ 1 (with the clarification that changes in alertness cannot be attributable to cerebral edema); 6.Meeting any of the following criteria:

1. ASPECTS 3-5 and NIHSS ≥ 30;
2. ASPECTS 0-2; 7.Signs on CT/MRI of an infarct of at least 50% of the middle cerebral artery territory; 8.No midline shift or midline shift <5mm; 9.Mechanical Thrombectomy and successful recanalization (defined as eTICI ≥2b50); 10.Ability to initiate decompressive hemicraniectomy within 6 hours after completion of mechanical thrombectomy and within 4 hours after randomization; 11.Informed consent obtained from the patient or his/her legal representative.

Exclusion Criteria:

Clinical Exclusion Criteria

1. Any symptoms and signs of brain herniation before randomization, such as pupil anisocoria and unstable vital signs.
2. In the judgment of the investigator, the subject is likely to have supportive care withdrawn in the first day.
3. Commitment to decompressive hemicraniectomy (DHC) prior to enrollment.
4. Severe, sustained hypertension (systolic blood pressure > 220 mm Hg or diastolic blood pressure > 110 mm Hg);
5. Baseline blood glucose <50 mg/dl (2.8 mmol/L) or >400 mg/dl (22.2 mmol/L);
6. Baseline platelet count <100 x10^9/L;
7. Known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with international normalized ratio > 1.7;
8. Severe renal insufficiency, defined as serum creatinine > 3.0 mg/dl (or 265.2 μmol/l) or glomerular filtration rate [GFR] < 30 ml/min, or patients requiring hemodialysis or peritoneal dialysis;
9. Patients that cannot complete 90-day follow-up (such as no fixed residence, overseas patients, etc.);
10. Suspected vasculitis or septic embolism;
11. Neurological diseases or mental disorders before onset that affect the assessment of the condition;
12. Females who are pregnant or in lactation;
13. Participating in other clinical trials that could confound the evaluation of the study;
14. Subjects who, in the opinion of the investigator, have a life expectancy <3 months due to conditions not related to current LHI or are unlikely to comply with follow-up requirements. Other conditions that the investigators believe are not suitable for participation or may pose a significant risk to the patient.

Neuroimaging Exclusion Criteria

1. Evidence of other brain diseases such as cerebral trauma, intracranial tumor (except small meningioma), cerebral aneurysm, etc.
2. Evidence of acute ischemic infarction in bilateral anterior circulation territory or involvement of posterior circulation territories (other than in patients with a fetal or near-fetal PCA configuration);
3. Vascular perforation during thrombectomy;
4. The pre-randomization CT findings exhibits evidence of parenchymal hemorrhage 2 intracranial hemorrhage, diffuse severe subarachnoid hemorrhage, or intraventricular hemorrhage. Patients with localized mild subarachnoid hemorrhage, hemorrhagic infarction type1 or 2, and small parenchymal hematoma type 1 without midline shift may be included;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-07-19 (Actual); Primary Completion 2029-06-19 (Estimated); Study Completion 2029-06-19 (Estimated)

PRIMARY OUTCOMES:
Rate of mRS score of 0-4 | 90 days (±7 days) after randomization
  Rate of mRS score of 0-4

SECONDARY OUTCOMES:
Rate of mRS score of 0-3 Ordinal shift analysis of mRS •Rate of mRS score of 0-2 •Rate of midline shift ≥ 5 mm •Rate of brain herniation Improvement of the NIHSS Rate of neurological deterioration Rate of rescue decompressive hemicraniectomy | 90 days (±7 days) after randomization
  mRS score ranges 0-6
Ordinal shift analysis of mRS | 90 days (±7 days) after randomization
  mRS score ranges 0-6
Rate of mRS score of 0-2 | 90 days (±7 days) after randomization
  mRS score ranges 0-6
Rate of midline shift ≥ 5 mm | Within 72 hours after randomization
  Based on imaging assessment (e.g., CT, MRI)
Rate of brain herniation | Within 72 hours after randomization
  e.g., 1 or 2 dilated, fixed pupils; unconsciousness related to edema [i.e., ≥2 on item 1a on the NIHSS]; and/or loss of other brain stem reflexes, attributable to edema or herniation according to the Investigator's judgment
Improvement of the NIHSS | 5-7 days after randomization or discharge
  The NIHSS score range from 0 (no deficit) to 42 (maximum deficit)
Rate of neurological deterioration | 5-7 days after randomization or discharge
  Defined as increase of NIHSS score ≥4 from baseline
Rate of rescue decompressive hemicraniectomy | 5-7 days after randomization or discharge
  Control group
Length of ICU stay | Perioperative
  Residual stay days of ICU
Length of hospitalization | Perioperative
  Residual stay days of hospitalization
Barthel Index | 90 days (±7 days) after randomization
  The Barthel Index range from 0 (severe disability) to 100 (no disability)
Modified Rankin scale and Barthel Index | 12 months (±30 days) after randomization
  The mRS score range from 0 (no disability) to 6 (death), the Barthel Index range from 0 (severe disability) to 100 (no disability)
Rate of any intracranial hemorrhage (ICH) | Within 72 hours after randomization
  The occurrence of ICH includes the following scenarios:
  1. new occurrence of ICH;
  2. progression of ICH based on Heidelberg Bleeding Classification.
Rate of parenchymal hematoma type 2 intracranial hemorrhage | Within 72 hours after randomization
Mortality | 90 days (±7 days) after randomization
  Defined as mRS 6
Serious Adverse Events | 90 days (±7 days) after randomization
  Detailled description noted in study protocol

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xuanwu Hospital, Capital Medical University., Beijing
  - Liaocheng Brain Hospital, Shandong